CLINICAL TRIAL: NCT05489367
Title: Does COVİD-19 m-RNA Vaccine Affect Fertility and Over Reserve ?
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Yıldız, DOCTOR, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasaTREHm
Record Dates: First submitted 2022-01-30; First posted 2022-08-05 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Virus Infection; Ovarian Function Insufficiency; Fertility Disorders; Vaccine Adverse Reaction
Keywords: ovarian reserve; covid-19; vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Pre-vaccine ovarian reserve and fertility status: Before vaccination, ovarian reserve tests and fertility status of 64 women will be examined and results will be recorded.After 2 doses of vaccination, ovarian reserve and fertility status of same 64 women will be examined and results will be recorded
  Interventions: Biological: sars cov 2 biontec vaccine

INTERVENTIONS:
Biological: sars cov 2 biontec vaccine — volunteers will be expected to receive 2 doses of vaccine

SUMMARY:
Women's ovarian reserve and fertility were compared before and after 2 doses of vaccination

DETAILED DESCRIPTION:
our study ıs desıgned as an observatıonal clınıcal study. the purpose ıs to compare the over reserve tests of the patıents before and after vaccıne, to determıne ıf the over reserve and fertılıty of women are affected by the vaccıne.women who applied to the vaccination outpatient clinic for the first dose of vaccine were included in the study.those who have never been vaccinated and have not had covid 19 infection were included in the study.antı ullerıan hormone level ıs the laboratory parameters that best showıng the ovary reserve today. ovarian reserve tests including amh were checked and their fertility was questioned and their information was recorded.

the same tests were repeated after the volunteers received 2 doses of vaccine. ın the power analysis, it was calculated that 104 volunteers should be included in the study.the study will be terminated when 104 volunteers are reached.

ELIGIBILITY:
Inclusion Criteria:

* between 18-45 years old
* have ever had a covid vaccine
* not be infected with covid 19

Exclusion Criteria:

* pregnancy
* diagnosis of any kind of cancer
* oral contraceptive usage
* endometrioma
* PCOS
* menopause
* menstrual irregularity
* premature ovarian insufficiency

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — volunteers with functional ovaries and female gender
Study Population: 74 ovulatory women who were not vaccinated with Biontech.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Ovarian reserve tests and fertility status of 74 women before and after vaccination | 6 months after receiving the 2nd dose of vaccine
  before and after vaccination serum Amh level ng/ml

SECONDARY OUTCOMES:
AMH difference between vaccinated and unvaccinated groups | 6 months
  AMH difference between vaccinated and unvaccinated groups

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
A number will be given to each volunteer who agrees to participate in the study.All data obtained will be recorded in this number and all data will be stored on the personal computer of the researcher.No personal data will be shared with anyone other than the study.